CLINICAL TRIAL: NCT06594848
Title: Investigating the Effects of Dietary Supplementation With a Black Rice Anthocyanidin Rich Extract (BRE) and Anthocyanidin Metabolites on the Synthesis and Release of Brain Derived Neurotropic Factor (BDNF) in Healthy Subjects
Brief Title: Effects of a Black Rice Extract and Anthocyanidin Metabolites on the Synthesis and Release of BDNF in Healthy Subjects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2186403
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cognition - Other; Depression, Anxiety
Keywords: Anthocyanin; cyanidin; BDNF; Metabolites
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo consists in 4 g of maltodextrin with food coloring (blue and green dyes) to match the color on the active comparator (Black Rice Extract). The placebo will be dissolved in 200 ml of water.
  Interventions: Other: Placebo
- Black rice extract (Active Comparator): Active comparator consists in 2 g of Black Rice Extract and 2 g of maltodextrin. The Black Rice Extract will be dissolved in 200 ml of water.
  Interventions: Dietary Supplement: Black rice extract

INTERVENTIONS:
Dietary Supplement: Black rice extract — Black rice extract is rich in a specific type of anthocyanins, cyanidin. It has been shown by our group that cyanidin-rich food can have beneficial health effects
  Arms: Black rice extract
Other: Placebo — The placebo for this study is composed by maltodextrin and food colorant
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effect of black rice extract (BRE) supplementation on levels of BDNF, which is a key molecule in cognition in healthy volunteers. The main questions to answer are:

Does single BRE consumption increase levels of BDNF in the circulation in healthy men and women? Does single BRE consumption impact BDNF gene expression in cells isolated from the blood?

Researchers will compare BRE to a placebo (a look-alike supplement that contains no BRE) to see if BRE increases levels of BDNF in blood.

DETAILED DESCRIPTION:
The first study will be a cross over-double blind placebo controlled, the second will be and ex vivo study.

Subjects will initially be pre-screened for eligibility by a phone interview to determine if they meet basic study inclusion and exclusion criteria and wish to proceed with the in-person screening. Interested subjects that meet both inclusion and exclusion criteria based on the phone interview will be invited to the Ragle Facility (Ragle Human Nutrition Research Center, Academic Surge II, UCD main campus) for an in-person screening visit. During this visit, the aim of the study the participant chooses to be in and how it will be conducted will be explained and written. Informed consent will be obtained from the potential participants.

For the first study, subjects will be asked for: i) being fasted for at least 12 h; ii) determination of body weight, height, and blood pressure; iii) a finger stick blood sample to determine actual glucose and triglyceride concentrations; and iv) answering a health and habits questionnaire. The responses to the questionnaire and the results from the screening measurements (BMI and blood pressure, blood glucose and triglycerides) will be used to confirm that potential participants meet inclusion/exclusion criteria.

For the second study, subjects will be asked for: i) being fasted for at least 12 h; ii) determination of body weight, height, and blood pressure; iii) a finger stick blood sample to determine actual glucose and triglyceride concentrations; and iv) answering a health and habits questionnaire. The responses to the questionnaire and the results from the screening measurements (BMI, blood pressure, blood glucose and triglycerides) will be used to confirm that potential participants meet inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is healthy and, in the opinion of the investigator, free of any medical conditions that might affect study measurements.
2. Male or female.
3. Age between 18 - 80 years inclusive.
4. BMI between 21 - 29.9 kg/m2.
5. Female subject of childbearing potential has a negative urine pregnancy test result.
6. Subject agrees to discontinue the use of pre- and/or probiotic and/or polyphenol supplements from 2 days prior to the screening and throughout the study.
7. Subject agrees to consume less than 1/2 cup/day of foods containing AC (such as blueberries, blackberries, bilberries, cherries, grapes, grape juice, pomegranate, raspberries, huckleberries, strawberries) and no more than 1 glass/day of red wine, 3 cups/day of tea or coffee, or 10 g/day of dark chocolate from 2 days prior to the screening and throughout the study.
8. No known allergies to study products or components (rice).
9. Subject is willing to consume a low fat/low flavonoid dinner the evening before study visits.
10. Subject has received a complete COVID-19 vaccine and is at least 6 weeks post-vaccine at the pre-screening visit as verified by shot record or similar documentation.
11. Subject has given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

1. Age < 18 or > 80 years.
2. BMI < 21 or > 29.9 kg/m2.
3. Vegan, Vegetarian, or other dietary restrictions that would not allow the subject to easily consume a low polyphenol diet leading up to screening and study visits.
4. Current consumption of special diets (e.g. Atkins, keto, paleo, etc.).
5. Current participation or enrollment in another pharmaceutical, weight-loss or nutritional clinical study within the last 30 days. Device trials are exempted.
6. Uncontrolled hypertension defined as diastolic blood pressure ≥ 95 mmHg and/or systolic blood pressure ≥ 160 mmHg.
7. Fasting blood triglycerides > 150 mg/dL.
8. Self-reported Type 2 Diabetes.
9. Fasting blood glucose <50 mg/dL or > 100 mg/dL.
10. Hemoglobin A1c levels ≥ 5.7%.
11. Current smoker or use of tobacco products within the last 180 days.
12. Binge drinking (alcohol intake ≥ 5 alcoholic drinks for males or ≥ 4 alcoholic drinks for females on the same occasion, i.e. at the same time or within a couple of hours of each other).
13. Substance abuse or dependence within the last 60 days.
14. Daily use of anti-inflammatory medications including NSAIDs and aspirin within the last 30 days.
15. Use of laxative medications or other products that promote colon cleansing within the last 30 days.
16. History of restricted diets or use of herbal supplements or medications that interfere with insulin metabolism within the last 30 days.
17. History of stroke, hepatic, gallbladder, kidney, thyroid disease, or cancer.
18. History of immune related disorders or Raynaud's disease.
19. Current clinically significant depression, anxiety, or other psychiatric condition.
20. History of malabsorption or GI tract disorders.
21. History of GI surgeries (e.g. lap band, gastric bypass, etc.).
22. Diarrhea or oral antibiotic intake within the last 30 days.
23. Weight change (> 5%) within the last 30 days.
24. History of eating disorders such as bulimia, anorexia, or muscle dysmorphia.
25. Allergy or sensitivity to the study products.
26. Subject has not received a complete COVID-19 vaccine or is less than 6 weeks post-vaccine at the screening visit.
27. Any other condition which in the Investigator's opinion might adversely affect the subject's ability to complete the study or its measurements or which might pose significant risk to the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
BDNF | Changes in circulating BDNF upon single consumption of black rice extract (4 hours kinetic)
  BDNF will be measured in the serum using ELISA kit following the manufacturers' instruction

SECONDARY OUTCOMES:
BDNF gene epxression in isolated blood cells | Changes in mRNA BDNF levels upon single consumption of black rice extract (4 hours kinetic)
  mRNA levels of BDNF will be measured using quantitative PCR

CONTACTS AND LOCATIONS:
Overall Officials: Eleonora Cremonini, Principal Investigator — UC Davis; Patricia I Oteiza, Principal Investigator — UC Davis
Locations (1):
- Ragle Human Nutrition Research Center, Academic Surge II, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No